CLINICAL TRIAL: NCT07397871
Title: Changes in Salivary Parameters in Patients Undergoing Clear Aligner Orthodontic Treatment: A Randomized Controlled Trial
Brief Title: Salivary Flow, pH, and Buffering Capacity in Fixed and Clear Aligner Orthodontic Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Omar Alkadhi, Associate Professor, Preventive Dentistry Department College of Medicine and Dentistry, Riyadh Elm University, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REU-CA-SALIVA-RCT-001
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Orthodontic Treatment; Saliva
Keywords: Salivary flow; Salivary pH; Buffering capacity; Fixed orthodontic appliance; Clear aligner therapy
MeSH Terms: interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: A non-inferiority randomized controlled trial with two parallel arms and an allocation ratio of 1:1.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor, and data analyst will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed orthodontic treatment control group (Active Comparator): Study subjects in control group will receive fixed orthodontic appliances with metallic brackets of 0.022-inch slot size (American Orthodontics). The bonding process will be performed using the same adhesive (BracePaste, American Orthodontics) for all patients, and treatment will be initiated with 0.014-inch NiTi archwires (Highland Metals).
  Interventions: Device: Fixed orthodontic appliances
- Clear Aligner Treatment Group (Experimental): Study subjects in Clear Aligner treatment group will receive Invisalign® (Align Technology, Inc., Tempe, AZ, USA). The Clear Aligner treatment protocol will be followed until the end of the treatment.
  Interventions: Device: Clear Aligner Treatment

INTERVENTIONS:
Device: Fixed orthodontic appliances — Study subjects in control group will receive fixed orthodontic appliances with metallic brackets of 0.022-inch slot size (American Orthodontics).
  Arms: Fixed orthodontic treatment control group
Device: Clear Aligner Treatment — Study subjects in Clear Aligner treatment group will receive Invisalign® (Align Technology, Inc., Tempe, AZ, USA). The Clear Aligner treatment protocol will be followed until the end of the treatment.
  Arms: Clear Aligner Treatment Group

SUMMARY:
Study Design: A randomized controlled trial with two parallel arms and an allocation ratio of 1:1.

Setting: The study will be conducted in the orthodontic department of Riyadh Elm University hospitals in Riyadh City, Saudi Arabia.

Participants: Patients undergoing fixed or clear aligner orthodontic treatment referred to REU dental hospital will be randomly allocated to either the clear aligner group or the fixed orthodontic appliance group.

Intervention: Prior to orthodontic treatment, all patients will receive phase I periodontal therapy and oral hygiene instructions. Fixed orthodontic appliances will be bonded using metallic brackets with a 0.022-inch slot and 0.014-inch NiTi archwires. Clear aligner patients will receive Invisalign® treatment.

Outcomes and Saliva Collection: Salivary samples will be collected using the spitting method at baseline (T0) and follow-up time points according to the study protocol. Salivary flow rate, pH, and buffering capacity will be assessed as described in the proposal.

Randomization and Blinding: Randomization will be performed using a random number generator with allocation concealment via opaque envelopes. The investigators involved in outcome assessment and data analysis will be blinded.

Ethical Considerations: The study will be submitted to the Institutional Review Board at Riyadh Elm University and conducted in accordance with IRB policies.

DETAILED DESCRIPTION:
This study is a randomized controlled clinical trial designed to evaluate changes in salivary parameters in patients undergoing fixed orthodontic treatment or clear aligner therapy. Patients referred to the orthodontic department of Riyadh Elm University dental hospital will be screened for eligibility and randomly allocated into two parallel groups with an allocation ratio of 1:1.

Prior to the initiation of orthodontic treatment, all participants will undergo phase I periodontal therapy and receive standardized oral hygiene instructions. Patients in the fixed orthodontic appliance group will be treated using metallic brackets with a 0.022-inch slot and initial 0.014-inch nickel-titanium archwires. Patients in the clear aligner group will receive clear aligner treatment according to the prescribed protocol.

Salivary samples will be collected using the spitting method at baseline before the start of orthodontic treatment (T0) and at subsequent follow-up time points as specified in the study protocol. Salivary flow rate, salivary pH, and buffering capacity will be assessed at each time point using standardized methods described in the proposal.

Randomization will be carried out using a random number generator, with allocation concealment ensured through the use of opaque sealed envelopes. The investigators involved in outcome assessment and data analysis will be blinded to group allocation.

This study will be conducted following approval from the Institutional Review Board (IRB) of Riyadh Elm University and in accordance with institutional ethical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Class I, II and III skeletal malocclusion.
* Age ≥18 undergoing fixed or Clear aligner orthodontic treatment.

Exclusion Criteria:

* Current medications including antibiotic use within the past 3 months that affect salivary flow and composition.
* Active smoking including vaping and E-cigarette use.
* Diagnosis of systemic diseases/conditions such as Sjogren's syndrome, diabetes, chronic kidney diseases, neurological conditions.
* Active dental caries or signs of gingivitis and/or periodontitis
* Less than three months of orthodontic treatment since it is characterized by acute, temporary changes and patient adaptation to the new appliances.
* Requiring single arch treatment to standardize the research and eliminate a potential confounding variable
* Crown restoration is excluded due to their material properties which may affect salivary composition.
* Pregnancy due to the physiological variation in salivary flow and composition due to hormonal changes.
* Presence of mouth breathing may lead to inconsistent salivary flow rate, Changes in Salivary Composition and pH
* Poor oral hygiene with high levels of dental plaque, calculus, and gingival inflammation can independently alter salivary flow rate, pH, and buffer capacity there by acting as confounding variable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-05-29 (Estimated)

PRIMARY OUTCOMES:
Salivary flow rate | The outcome measure will be assessed at (T0) just before the commencement of fixed appliance and Clear Aligner therapy, at one week (T1), at two weeks (T2), after three months (T3), and at six months (T4) of treatment.
  The salivary flow rate will be recorded in each patient. Two mL of whole unstimulated saliva will be collected in a graduated tube. The salivary flow rate will be recorded in all the four time points T0, T1, T3 and T4.

SECONDARY OUTCOMES:
Salivary pH | The outcome measure will be assessed at (T0) just before the commencement of fixed appliance and Clear Aligner therapy, at one week (T1), at two weeks (T2), after three months (T3), and at six months (T4) of treatment.
  The pH values will be assessed using portable pH meter strips at the same four time points. Salivary pH will be measured at T0, T1, T3 and T4.
Salivary buffering capacity | The outcome measure will be assessed at (T0) just before the commencement of fixed appliance and Clear Aligner therapy, at one week (T1), at two weeks (T2), after three months (T3), and at six months (T4) of treatment.
  Buffer capacity will be determined by quantitative test using a hand-held pH meter method. This method will involve addition of 0.5 ml of saliva to 1.5 ml of 5 mmol/L HCl. Mixtures will be vigorously shaken. Then stream of Nitrogen will be passed through the mixture for 20 min to eliminate carbon dioxide from the sample and allowed to stand for 10 min when the final pH will be measured. The salivary buffering capacity will be measured at T0, T1, T3 and T4.

CONTACTS AND LOCATIONS:
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Romero G. [Therapeutic study of the use of Bay 2502 in young adults with chronic Chagas' infection]. Bol Chil Parasitol. 1969 Jan-Mar;24(1):97-9. No abstract available. Spanish. PMID 4983561
- [Background] Leone CW, Oppenheim FG. Physical and chemical aspects of saliva as indicators of risk for dental caries in humans. J Dent Educ. 2001 Oct;65(10):1054-62. PMID 11699977
- [Background] Alshahrani I, Hameed MS, Syed S, Amanullah M, Togoo RA, Kaleem S. Changes in essential salivary parameters in patients undergoing fixed orthodontic treatment: A longitudinal study. Niger J Clin Pract. 2019 May;22(5):707-712. doi: 10.4103/njcp.njcp_606_18. PMID 31089027
- See also: Arab S, Nouhzadeh Malekshah S, Abouei Mehrizi E, et al. (2016) Effect of Fixed Orthodontic Treatment on Salivary Flow, pH and Microbial Count. Journal of Dentistry (Tehran, Iran) 13(1): 18-22. Razan'S Alsalamah Proposal 3-To… — https://pmc.ncbi.nlm.nih.gov/articles/PMC4983561/
- See also: Dawes C (2003) What is the critical pH and why does a tooth dissolve in acid? Journal (Canadian Dental Association) 69(11): 722-724. — https://pubmed.ncbi.nlm.nih.gov/14653937/
- See also: Leone CW and Oppenheim FG (2001) Physical and chemical aspects of saliva as indicators of risk for dental caries in humans. Journal of Dental Education 65(10): 1054-1062. — https://pubmed.ncbi.nlm.nih.gov/11699977/